CLINICAL TRIAL: NCT02399254
Title: The Trajectory of Physical Activity Following Pulmonary Rehabilitation
Status: Completed | Type: Observational
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Other Study IDs: 14-06-001 E
Record Dates: First submitted 2015-03-16; First posted 2015-03-26 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-04

CONDITIONS: COPD; Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary Rehabilitation: Chronic Obstructive Pulmonary Disease (COPD) patients following pulmonary rehabilitation

SUMMARY:
Pulmonary rehabilitation clearly increases exercise capacity, but its effect on physical activity in the home and community settings is less clear. It may take a longer time for this increase in physical activity to occur. It has been stated in an editorial that it takes 3 months to train the muscles but 6 months to train the brain. The Investigators will first evaluate the change in physical activity following pulmonary rehabilitation using state-of-the-science motion detectors, then Investigators will follow the trajectory of physical activity over the next several months.

DETAILED DESCRIPTION:
This study will follow physical activity following pulmonary rehabilitation longitudinally over 48 weeks. Investigators will use a state-of-the-art accelerometer, to analyze minutes walking per day as the primary outcome, rather than vector magnitude units (VMU) or estimated steps per day. Investigators will explore potential factors influencing this important outcome, including baseline activity levels, demographic variables, changes in exercise capacity, psychological variables, and self-efficacy scores. Finally, Investigators will evaluate the rate of change (trajectory) in physical activity over approximately six months after pulmonary rehabilitation. There are limited data suggesting it takes time for the translation of increased exercise capacity into increased physical activity to occur.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 40 years) with a primary clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
2. A post-bronchodilator forced expiratory volume in one second(FEV1)/forced vital capacity (FVC) < 0.70 from spirometry performed within the preceding 12 months (no specific FEV1 percent-predicted requirement, although we anticipate the FEV1 will average around 45% of predicted, based on previous studies of pulmonary rehabilitation)
3. The patient was referred to pulmonary rehabilitation
4. The patient is clinically-stable: no exacerbation in preceding 4 weeks
5. Modified Medical Research Council (mMRC) dyspnea rating of at least 2 out of 5.

Exclusion Criteria:

1. Disease severity or co-morbidity that would make the patient be at-risk for participation this study
2. A significant movement disorder, such as hemiplegia, etc.
3. Inability to read and comprehend the questionnaires, which will be in English
4. A history of poor wound healing or chronic skin conditions that might predispose to local problems from wearing the DynaPort. (The DynaPort can be worn outside a thin garment, such as a tee shirt, and is relatively thin, without protruding parts. However, since the device may be worn overnight, and there is a remote risk of pressure problems, this exclusion criterion was added).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary Rehabilitation Center
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-04; Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard ZuWallack, MD, Principal Investigator — Saint Francis Hospital and Medical Center
Locations (4):
- United States (4):
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Gaylord Hospital, Wallingford, Connecticut
  - VA Connecticut Research and Education Foundation, West Haven, Connecticut
  - Ocean State Research Institute, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulmonary Rehabilitation: COPD patients following pulmonary rehabilitation
Period: Overall Study
Arm/Group | Pulmonary Rehabilitation
Started | 21
Completed (Transferring activity data was an issue at all sites despite good support from the manufacturer.) | 19
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Minutes/Day at 12 Weeks
Description: Investigators will look at changes in directly-measured physical activity (minutes per day of walking activity from the DynaPort) between the 12 ± 3 week assessment and baseline.
Time Frame: 12 weeks compared to baseline
Population: Obtaining valid activity data (uploaded to the manufacturer then downloaded to the site) was a problem at all sites despite good support from the manufacturer. As a result a N of 16 could be analyzed at week 12.
Measure: Mean (Standard Error); unit: minutes/day
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 16
minutes/day | 1.3125000 (0.7400380)

2. Primary Outcome: Minutes/Day at 48 Weeks
Description: Investigators will look at changes in directly-measured physical activity (minutes per day of walking activity from the DynaPort) between the 48 ± 3 week assessment and baseline.
Time Frame: 48 weeks compared to baseline
Population: Obtaining valid activity data (uploaded to the manufacturer then downloaded to the site) was a problem at all sites despite good support from the manufacturer. As a result a N of 10 could be analyzed at week 48.
Measure: Mean (Standard Error); unit: minutes/day
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 10
minutes/day | 0.5000000 (1.0979779)

3. Secondary Outcome: Activity-related Energy Expenditure (AEE)(J/Min/kg) at 12 Weeks
Description: Investigators will look at changes in activity-related energy expenditure (from the DynaPort) at 12 weeks compared to baseline
Time Frame: 12 weeks compared to baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: AEE (J/min/kg)
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 16
AEE (J/min/kg) | 4.9375000 (1.9737206)

4. Secondary Outcome: Activity-related Energy Expenditure (AEE)(J/Min/kg) at 48 Weeks
Description: Investigators will look at changes in activity-related energy expenditure (from the DynaPort) at 48 weeks compared to baseline
Time Frame: 48 weeks compared to baseline
Population: as for outcome 2
Measure: Mean (Standard Error); unit: AEE (J/min/kg)
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 10
AEE (J/min/kg) | 2.9000000 (1.9405039)

ADVERSE EVENTS:
Time Frame: 48 Weeks
Description: Events reported by subjects at 12 week visit 24 week visit,36 week visit and 48 week visit
Arm/Group | Pulmonary Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 10/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulmonary Rehabilitation (N=21)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 7 (9) — Chronic obstructive pulmonary disease exacerbation,Shortness of breath
Diarrhea (Gastrointestinal disorders) | 1 (1) — Loose bowel, loose stools
Pneumonia (Infections and infestations) | 1 (1)
Cholelithiasis (General disorders) | 1 (1) — gallstones, gall bladder stones
Deep Vein Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT02399254/Prot_SAP_000.pdf